CLINICAL TRIAL: NCT06780852
Title: A Pilot Clinical Study to Evidence Improved Cranial Flap Fixation With a Bioresorbable Bone Adhesive Based on Imaging and Patient Reported Outcomes
Brief Title: A Pilot Clinical Study to Evidence Improved Cranial Flap Fixation With a Bioresorbable Bone Adhesive
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RevBio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DVAL22023
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Craniotomy
Keywords: cranial flap fixation; bone adhesive; bioresorbable

STUDY DESIGN:
Intervention Model Description: This will be a single-center, two-arm, prospective study in which 15 qualified patients in need of a cranial flap fixation following a craniotomy will be enrolled. To begin the study, 5 patients will undergo cranial flap fixation using currently. marketed hardware (standard of care), with TN-CFF used to augment the fixation hardware and fill the kerf line. After the completion of the first 5 patients, 10 patients will undergo cranial flap fixation using only Tetranite for Cranial Flap Fixation (TN-CFF).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Hardware Augmentation (Experimental): The first 5 patients will undergo cranial flap placement using currently marketed metal fixation (plates and screws). The kerf line and burr holes will then be filled with Tetranite (TN-CFF).
  Interventions: Device: Tetranite for Cranial Flap Fixation (TN-CFF)
- Standalone (Experimental): The patients will undergo cranial flap fixation using only Tetranite (TN-CFF) for Cranial Flap Fixation.
  Interventions: Device: Tetranite for Cranial Flap Fixation (TN-CFF)

INTERVENTIONS:
Device: Tetranite for Cranial Flap Fixation (TN-CFF) — Bioresorbable bone adhesive for cranial flap fixation following a craniotomy.

SUMMARY:
This clinical pilot study will evaluate the use of a bioresorbable bone adhesive to improve cranial flap fixation at two study time points (at the time of fixation and 6 months). The aim of this Pilot Study is to demonstrate the safety and efficacy of the use of Tetranite for Cranial Flap Fixation (TN-CFF) to allow clinical study of the TN-CFF device in a greater number of patients.

DETAILED DESCRIPTION:
The primary endpoint is safety during the post procedure follow up period. This endpoint will be evaluated through the rate of all serious adverse device and procedure related effects from the time of fixation to 6 months post-procedure. The secondary endpoints include efficacy evaluated through radiolucency data using CT imaging at the cranial flap cut lines and the change of radiolucency with respect to time, device related adverse events, flap immobility at time of fixation, six months and 12 months, evaluation of flap translation and patient reported outcome measures.

ELIGIBILITY:
Inclusion Criteria:

Subjects or representatives must have voluntarily signed the informed consent form before any study related procedures;

* Subjects can be any gender, but be between (and including) 18 and 75 years of age
* Subject is scheduled for a cranial procedure in the supratentorial location.
* Subject requires a procedure involving a Class I/clean wound (uninfected surgical wound in which no inflammation was encountered).
* Subject, and/or subject's family are able and willing to provide informed consent and HIPAA authorization.
* Subject is able and willing to meet all study requirements, including attending all post-index procedure assessment visits and radiological tests.

Intra-Operative Inclusion Criteria:

* Width of craniotomy kerf line < 3mm for more than 75% of the bone flap border

Exclusion Criteria:

* Subject requires a procedure involving a translabyrinthine, transsphenoidal, transoral approach, or any procedure that penetrates the air sinus or mastoid air cells. Note: Superficial penetration of mastoid air cells is not an exclusion if cells were appropriately sealed (e.g., bone wax).
* Subject has clinically significant hydrocephalus or clinical evidence of altered CSF dynamics.
* Subject has undergone a previous, open intracranial neurosurgical procedure in the same anatomical location. (Note: stereotactic biopsy was not exclusionary).
* Subject requires a craniectomy (the bone flap is not replaced during the current surgery).
* Subject had radiation treatment to the surgical site, or standard fractionated radiation therapy was planned post index-procedure. (Note: stereotactic radiosurgery prior to the planned index procedure was not an exclusion criterion.)
* Subject requires a craniotomy across the sinus for which Tetranite is applied adjacent to or within the sinus to fixate the cranial flap.
* Subject has a condition with anticipated survival shorter than six months.
* Subject has undergone chemotherapy treatment, excluding hormonal therapy, within three weeks prior to the planned index procedure, or use of intracavitary chemotherapy wafer (BCNU) was planned, or chemotherapy treatment was planned within two weeks after the index procedure was performed.
* Standard use of peri-operative steroids (i.e., corticosteroids) is permitted. Chronic steroid use (defined as daily use of corticosteroids for ≥ 8 weeks) for the purposes of reducing the side effects of chemotherapy and/or radiation therapy for cancer is not exclusionary unless the patient is deemed by the investigator to be suffering from steroid toxicity (i.e., Cushing's syndrome) manifested by symptoms and signs such as thin skin, striae, easy bruising, muscle atrophy, upper body obesity, severe fatigue, etc. Use of corticosteroids on a chronic basis (as defined previously) for purposes other than decreasing the symptoms of systemic chemotherapy is exclusionary unless those steroids were discontinued 4 weeks prior to the planned index procedure.
* Subject receives warfarin, heparin, other anticoagulant agents on a daily basis and pre-surgical, standard of care drug wash-out did not occur.
* Subject is pregnant, breast-feeding, or intended to become pregnant during the course of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the rate of all serious adverse device and procedure related effects during the post procedure follow up period. | Time of fixation and 6 months post-procedure.
  Rate of all serious adverse device and procedure related effects from the time of fixation to 6 months post - procedure

SECONDARY OUTCOMES:
Radiolucency data using CT imaging at the cranial flap cut lines. | Throughout 12 Months post-procedure period.
  Radiolucency data using CT imaging at the cranial flap cut lines and the change of radiolucency with respect to time.
Device-related adverse events | Throughout 12 Months post-procedure period.
  Device-related adverse events included all adverse events classified as definitely, probably, possibly, or undetermined relation to the device or procedure.
Flap immobility determined clinical palpation of the cranial flap by an independent neurosurgeon. | Time of fixation and 6 months post-procedure.
  Flap immobility will be determined by an independent neurosurgeon.
Flap immobility as determined by clinical palpation of the cranial flap by the neurosurgeon and the patient. | 6 months and 12 months post-procedure.
  Flap immobility will be determined by the surgeon and the patient.
Translation of the flap based on CT scan. | Throughout 12 Months post-procedure period.
  Translation of the flap based on CT scan
Patient Reported outcome using PROMIS10 | Throughout 12 Months post-procedure period.
  Subject satisfaction after TN-CFF was used for cranial flap fixation using a validated questionnaire for overall health.
Patient Reported outcome using the 36 Item Short Form Survey (SF-36). | Throughout 12 Months post-procedure period.
  Subject satisfaction after TN-CFF was used for cranial flap fixation using a validated questionnaire for overall quality of life measures.
Patient Reported outcome as measured on a Visual Analog Scale of pain intensity. | Throughout 12 Months post-procedure period.
  Subject satisfaction after TN-CFF is used for cranial flap fixation (i.e., level of headache pain)

OTHER OUTCOMES:
Neurological Exam using the Karnofsky Performance Scale (KPS) | Throughout 12 Months post-procedure period.
  Neurological exam will be completed throughout the study to assess neurological healing. The KPS scale is designed to measure the level of patient activity and medical care requirements
Neurological Exam using the Neurologic Assessment in Neuro-Oncology (NANO) scale. | Throughout 12 Months post-procedure period.
  Neurological exams will be completed throughout the study to assess neurological healing. The NANO scale is a quantifiable evaluation of 9 relevant neurologic domains based on direct observation and testing conducted during routine office visits.
Wound Healing | Throughout 12 Months post-procedure period
  Wound healing will be evaluated at post-surgical visits and will result in one of the three results: Surgical Revision needed, Superficial dehiscence, Completely Healed
Patient reported outcomes will also be measured using a patient taken picture of surgical wound. | Throughout 12 Months post-procedure period.
  A patient taken picture of surgical wound will be taken to show wound progress.
Patient Reported Outcome using a Cranio-facial assessment survey. | Throughout 12 Months post-procedure period.
  Subject satisfaction after TN-CFF was used for cranial flap fixation using a questionnaire for overall quality of life measures.
Qualitative assessment of artifact and distortion of MRIs. | Throughout 12 Months post-procedure period.
  Assessment of artifact and distortion on MRIs (for cases when imaging is available)

CONTACTS AND LOCATIONS:
Overall Officials: Kumar Abhinav, BSc MBBS MD FRCS(Neurosurgery), Principal Investigator — Bristol Southmead Hospital
Locations (1):
- Bristol Southmead Hospital, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD at this time. Study results will be published in a journal after study completion.